CLINICAL TRIAL: NCT00928941
Title: Neural Correlates of Cognitive Rehabilitation in PTSD
Brief Title: Neural Correlates of Cognitive Rehabilitation in Post-Traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left the project and the VA, as of 3/2011
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B7009-M; B7009-M (Other Grant/Funding Number: VA RR&D); NCT01584349 (obsolete NCT alias)
Record Dates: First submitted 2009-06-22; First posted 2009-06-26 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; rehabilitation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): A cognitive training program (Posit Science) or an active control (video game) will be implemented for at least 3-4 hours a week for 40 training units.
  Interventions: Behavioral: cognitive training
- Arm 2 (Active Comparator): A computer game control condition will be implemented for 3-4 training exercises a week for 40 hours.
  Interventions: Behavioral: video game

INTERVENTIONS:
Behavioral: cognitive training — A cognitive training program (Posit Science) or an active control (video game) will be implemented for at least 3-4 hours a week for 40 training units/hours.
  Arms: Arm 1
Behavioral: video game — An active control condition (computer game without increasing difficulty) will be implemented for at least 3-4 hours a week for 40 hours.
  Arms: Arm 2

SUMMARY:
Post Traumatic Stress Disorder (PTSD) is an emotional disorder that can also lead to problems with attention and memory. Cognitive training has been successfully used to improve attention and processing speed in other patient populations as well as healthy elderly. The purpose of this study is to examine how effective cognitive training will be in Veterans with PTSD.

DETAILED DESCRIPTION:
1. Objective(s) Post Traumatic Stress Disorder (PTSD) has been established as relatively common in a significant number of OEF/OIF Veterans (Vasterling & Brailey, 2005; Hoge et al., 2008). Attention deficits, which are prominent in PTSD, may be due to difficulty sustaining attention over time and encoding or getting information into storage which leads to reduced attention and memory scores on neuropsychological measures. Disruptions in attention are common in many types of neurological and psychiatric disorders. Deficient attentional skills may negatively affect cognitive performance in other areas (e.g., memory, planning) and thereby reduce effectiveness navigating daily life tasks as well as decrease the Veteran's life satisfaction after returning home.

   The origin of the attention impairment may be amenable to sophisticated remediation approaches using a "bottom up, neuroscience based" visual training program (i.e., Posit Science, Inc. cognitive rehabilitation program), which has been successful in improving neurocognitive function in healthy older adults (e.g., Mahncke et al., 2006) and patients with Schizophrenia (e.g., Bell at al., 2008). By engaging Veterans with PTSD in targeted remediation, it is expected that both behavioral (seen in neuropsychological test gains) and neural activity (e.g., BOLD response through fMRI) will reflect the improvement and this may be linked to improved outcomes in daily functioning.
2. Research Design: The longitudinal research design for this project will be a three factor mixed factorial design with between subject factors of PTSD (+PTSD x -PTSD) and cognitive remediation [cogrem x video game] and within subject variable of time tested (pre-training, post-training, 3 month follow up). There will be 40 participants enrolled in the following groups of 10 each: 1) +PTSD/cogrem, 2) +PTSD/video game, 3) -PTSD/cogrem, and 4) -PTSD/video game. PTSD status is determined by a diagnosis of PTSD identified through a clinical interview for DSM-IV diagnostic criteria for PTSD. The active treatment is cognitive training. Veterans in this group will receive the Posit Science (Mahncke et al., 2006) visual cognitive remediation paradigm of 40 hours of training. The control treatment is a video game designed by Nintendo for the DS handheld system, which intended to improve mental functioning called Brain Age (Nintendo, Inc.) which will be played for 40 hours. Groups will be compared on the difference scores for neuropsychological, neurobehavioral and neuroimaging data to see if there is a benefit in cognitive training and if that benefit is greater in the group with PTSD.
3. Methodology: Forty outpatient Veterans will be enrolled. All individuals will receive a neurobehavioral interview, neuropsychological testing and neuroimaging at the baseline visit, post training and at follow-up visits. After the baseline visit, each volunteer will be randomized to one of two conditions.
4. Findings: This is a new study and there are no findings to date.
5. Clinical Relationships: This study will examine the effects of a standard cognitive rehabilitation program with OEF/OIF veterans who have cognitive deficits due to PTSD.
6. This project will impact veterans' healthcare by identifying cognitive problems in PTSD and will test the ability of a rehabilitation program to remediate those problems.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF Veteran,
* meets DSM-IV criteria for PTSD,
* control group does not meet criteria for PTSD

Exclusion Criteria:

* prior history of significant head injury (LOC > 30 minutes) or other neurological disorder (e.g., stroke, seizure, multiple sclerosis), learning disability or confirmed diagnosis of ADHD,
* contraindication to MR imaging, failed malingering tests during testing, or a history of severe mental illness (i.e., Schizophrenia, Bipolar Disorder)
* individuals will be excluded if in the 30 days prior to the initial interview if they:

  * do not have stable housing (i.e., staying in same residence),
  * have medication changes or have had a psychiatric hospitalization,
* participants who meet DSM-IV criteria for substance dependence will be excluded from the study,
* individuals will also receive urine toxicology and Breathalyzer testing as the first procedure on the evaluation day (pre and post treatment and at 3 month follow up); participants who test positive for alcohol or recent substance use (e.g., methamphetamine) or report significant levels of drug or alcohol use if they are unable to abstain from substance use at three consecutive visits
* veterans who are currently engaged in therapy treatment for PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
neuropsychological test data | post-training and 3 month follow up

SECONDARY OUTCOMES:
MRI data | post-training and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Wrocklage, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States